CLINICAL TRIAL: NCT00003654
Title: Diagnostic Study of Patent Blue V Dye to Identify Sentinel Lymph Nodes in Patients With Stage I or IIA Breast Cancer
Brief Title: Diagnostic Study to Identify Sentinel Lymph Nodes in Women With Stage I or Stage II Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Purpose: Diagnostic
Other Study IDs: CDR0000066746; FRE-FNCLCC-96008; EU-98055
Record Dates: First submitted 1999-11-01; First posted 2004-08-26 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — iso-sulfan blue; Sentinel Lymph Node Biopsy; Technetium Tc 99m Sulfur Colloid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: patent blue V dye
Procedure: lymphangiography
Procedure: radionuclide imaging
Procedure: sentinel lymph node biopsy
Radiation: technetium Tc 99m sulfur colloid

SUMMARY:
RATIONALE: Diagnostic procedures, such as blue dye or imaging to identify sentinel lymph nodes, may improve the ability to detect the extent of disease and help plan effective surgery for removing breast tumors.

PURPOSE: Diagnostic trial to study the effectiveness of blue dye and an imaging procedure to identify the sentinel lymph node under the arm in women with stage I or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether the concept of a sentinel lymph node within the axillary nodal basin is valid in staging breast cancer. II. Determine the sensitivity of combined methods of identification of sentinel lymph nodes by patent blue V dye and gamma probe detection in these women.

OUTLINE: Patients receive patent blue V dye injection peritumorally prior to surgery. Preoperative lymphoscintigraphy is performed using technetium Tc 99 sulfur rhenium colloid injected around the tumor associated with intraoperative gamma probe detection. Nonpalpable tumors receive a localized injection using stereotactic injection techniques. Patients then undergo standard axillary (level I and II) lymph node dissection.

PROJECTED ACCRUAL: A total of 200 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven stage I or IIA invasive breast cancer T0, T1, or T2 (no greater than 3 cm), N0 Noninflammatory Nonmetastatic No ductal carcinoma in situ Eligible for breast-conserving surgery Hormone receptor status: Positive or negative

PATIENT CHARACTERISTICS: Age: Any age Sex: Female Menopausal status: Pre- and postmenopausal Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Not pregnant No allergy or sensitivity to radiopharmaceuticals or patent blue V dye

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy Chemotherapy: No prior neoadjuvant chemotherapy Endocrine therapy: No prior endocrine therapy Radiotherapy: No prior neoadjuvant radiotherapy Surgery: No prior breast surgical biopsy or axillary surgery

Ages: 0 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 1997-09 (Actual); Primary Completion 2000-01 (Actual); Study Completion 2000-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Rodier, MD, Study Chair — Centre Paul Strauss
Locations (1):
- Centre Paul Strauss, Strasbourg, France